CLINICAL TRIAL: NCT06709690
Title: A Fast, Quiet, Artificial Intelligence-based PET/MR Solution for Paediatric Diseases
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RuijinH 2024-467
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Paediatric Patients
Keywords: 18F-FDG PET/MR; pediatric; silent scan; flexible coil; deep learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric patients: Children who have clinical symptoms and are suspected of having malignant tumors after being evaluated by clinical pediatricians and require 18F-FDG PET/MR examination to further clarify their conditions.

SUMMARY:
To investigate the feasibility of deep learning-assisted rapid silent PET/MR in pediatric applications.

DETAILED DESCRIPTION:
This study aims to address the challenges faced by PET/MR in pediatric applications by leveraging new technologies such as flexible coils, silent sequences, and deep learning-based image reconstruction. The objective is to provide a rapid, silent, comfortable, and half-dose PET/MR imaging solution for pediatric patients, and to demonstrate its feasibility in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Children who have clinical symptoms and are suspected of having malignant tumors after being evaluated by clinical pediatricians and require 18F-FDG PET/MR examination to further clarify their conditions.
2. Signed and dated informed consent form
3. Commit to complying with the research procedures and cooperate in the implementation of the entire research process.
4. No gender restriction, aged between 0 and 18 years old.

Exclusion Criteria:

1. Patients with serious illnesses that researchers consider unsuitable for participation in this clinical study. Such as severe heart and lung failure, severe bone marrow suppression, severe liver and kidney dysfunction, etc.
2. Patients with severe claustrophobia，epileptic seizures, respiratory distress who cannot lie down, and patients with mental anomalies who are unable to cooperate.
3. Patients with metal implants such as pacemakers, artificial metal heart valves, and neurostimulators in their bodies.
4. Non-compliant person.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inpatients and outpatients at Ruijin Hospital who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lesion detection rate | 1 year
  Routine laboratory or imaging tests or pathology are performed based on clinical needs to assess the accuracy, sensitivity and specificity of rapid silent 18F-FDG PET/MR for lesion detection.
Completion of PET/MR examinations | 1 year
  Upon completion of the examination, record the rate of completion
Sedation during PET/MR examinations | 1 year
  Upon completion of the examination, record the rate of sedation and rate of secondary sedation
Qualitative image quality | 1 year
  Two experienced nuclear medicine physicians evaluated the overall quality of the images using a Likert 5-point scale for both the new imaging PET/MR protocol and the traditional imaging protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- China, Shanghai Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No